CLINICAL TRIAL: NCT06199687
Title: Use of Virtual Reality in Providing Pain Management, Comfort and Satisfaction After Thyroid-Parathyroid Surgery
Brief Title: Effect of Virtual Reality on Pain, Comfort and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sacide Yildizeli Topcu, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TUTF-GOBAEK 2022/300
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative; Patient Comfort; Patient Satisfaction; Thyroidectomy; Nursing
Keywords: Postoperative pain; Nursing care; Patient Comfort; Patient satisfaction; Virtual reality
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Experimental - Randomised Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients in the experimental group were shown a virtual reality video called 'Turkey 4K - Scenic Relaxation Film With Calming Music', containing images of nature and sea with music, for 15 minutes using virtual reality glasses.
  Interventions: Other: Use of Virtual Reality
- Control Group (No Intervention): Patients received standard care.

INTERVENTIONS:
Other: Use of Virtual Reality — Use of Virtual Reality after After Thyroid-Parathyroid Surgery
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to examine the effect of virtual reality application on pain management, comfort, and care satisfaction in patients undergoing thyroidectomy-parathyroidectomy. The main questions it aims to answer are:

1. Does the use of virtual reality reduce the level of postoperative pain in patients undergoing thyroid and parathyroid surgery?
2. Does the use of virtual reality increase the postoperative comfort level in patients undergoing thyroid and parathyroid surgery?
3. Does the use of virtual reality increase the level of satisfaction after surgery in patients undergoing thyroid and parathyroid surgery? Participants in the experimental group watched a virtual reality video containing nature and sea images and music playing in the background for 15 minutes. Participants in the control group received routine clinical care after thyroidectomy and parathyroidectomy. The pain levels of the patients in the experimental group were lower, and the comfort level was higher than in the control group. There was no difference between the groups in terms of satisfaction level with nursing care.

DETAILED DESCRIPTION:
Aim:

To examine the effect of virtual reality application on pain management, comfort and care satisfaction in patients undergoing thyroidectomy-parathyroidectomy.

Methods:

Settings and Design: This randomized controlled experimental study was conducted between February 6 - September 13 2023 with the participation of 69 patients who underwent thyroidectomy or parathyroidectomy in the general surgery unit of a university hospital.

The patients who underwent elective thyroidectomy or parathyroidectomy, had a postoperative drain, received the same analgesic treatment, stood up and started to feed orally, and agreed to watch videos with virtual reality glasses were included in the study.

Patients who have hearing problems and cannot speak Turkish and developed complications during the pre-operative and post-operative periods, who were diagnosed with severe visual impairment, epilepsy, and/or vertigo, and who experienced dizziness, nausea, and vomiting during the virtual reality application, were excluded from the study.

During the follow-up period of the study, one patient was excluded from the study because she experienced dizziness during the virtual reality application.

"Data Collection Form" was used to collect research data, "Numerical Evaluation Scale (0-10)" was used to evaluate the criteria regarding postoperative pain and satisfaction levels with nursing care, and "General Comfort Scale-Short Form" was used to evaluate the comfort criterion.

In order to avoid bias when grouping the patients to be included in the study, a randomization list was drawn up and the patients were randomly divided into 35 experimental groups and 35 control groups according to the order of hospitalization. In the randomization list made using the computer program, the letter "A" represented the experimental group and the letter "B" represented the control group.

During the data collection process, 70 patients who met the research criteria were interviewed and the patients were divided into two groups: the experimental group (35 patients) and the control group (35 patients). The randomization list was used to assign patients to groups. The experimental group consisted of patients who received postoperative virtual reality application, and the control group consisted of patients who received routine postoperative care. One patient in the experimental group was excluded from the study because he experienced dizziness during virtual reality application. The study was completed with 69 patients, 34 patients included in the experimental group and 35 patients assigned to the control group.

All patients received standard care after thyroid and/or parathyroid surgery. The standard care provided to the patients included nonsteroidal analgesic and antibiotic treatment administered twice a day (10:00, 22:00), as well as treatments and care to reduce sore throat and difficulty swallowing. In addition to receiving standard treatment and care, patients in the experimental group were allowed to watch virtual reality videos.

Patients who met the inclusion criteria for the study were visited in their rooms the day after the surgery (day 1 after surgery), at a time outside the clinic visit, meal, treatment and visiting hours. The patients were informed about the research and their written and verbal consent to participate in the study was obtained. All patients who agreed to participate in the study were asked by the researchers about their pain levels according to the questions in the data collection form and the numerical rating scale, and their answers were recorded.

In the experimental group, after recording the answers of the patients to the questions in the data collection form, a video called "Turkey 4K - Scenic Relaxation Film With Calming Music", containing nature and sea images with music was showed for 15 minutes with virtual reality glasses. Virtual reality glasses were disinfected after use for each patient. The patients' pain levels were re-evaluated after the virtual reality application was completed. Following the second pain assessment of the patients, evaluations were made regarding their comfort and satisfaction levels.

Pain levels of the patients who were in the control group were evaluated after recording their answers to the questions in the data collection form. After this evaluation, no intervention was made to the patients. After 15 minutes, the patients' pain intensity was re-evaluated and their comfort and satisfaction levels were also evaluated.

Pain evaluations of patients in both experimental and control groups were made between the 3rd and 4th hours following the last analgesic application. Patients in the experimental group were informed in detail about the use of virtual reality glasses before pain assessment, and their compliance with the virtual reality application was evaluated during the intervention. In the experimental group, it was observed that all patients adapted sufficiently to the application, except for one patient who experienced dizziness during the application. The data collection and application processes of the study took approximately 60 minutes for each patient.

Statistical Analysis Data obtained from 69 patients were analyzed using the IBM Statistical Package for the Social Sciences (SPSS) 22.0 (IBM, Armonk, New York, USA) package program. Normal distribution was determined by the Kolmogorov-Smirnov test. The Independent Sample t-Test was used to compare the pain, comfort and satisfaction scores between the two groups. Paired Sample t-Test was used to compare the means of pain, comfort and satisfaction scores scores within the group. The statistical significance level was accepted as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Underwent elective thyroidectomy or parathyroidectomy, Had a postoperative drain, Received the same analgesic treatment, Stood up and started to feed orally, Agreed to watch videos with virtual reality glasses

Exclusion Criteria:

Have hearing problems Can not speak Turkish Developed complications during the surgical process, Diagnosed with severe visual impairment, epilepsy, and/or vertigo, Experienced dizziness, nausea, and vomiting during the virtual reality application

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after virtual reality | Change in postoperative pain at the 15th minute after the virtual reality video ends
  Assessment of pain after watching a virtual reality video by using numerical pain scale (0-10)

SECONDARY OUTCOMES:
Patient comfort | Within 30 minutes after the virtual reality video ends
  Assessment of postoperative patient comfort after watching a virtual reality video
Patients satisfaction with nursing care | Within 30 minutes after the virtual reality video ends
  Assessment of patient satisfaction after watching a virtual reality video by using numerical pain scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Sacide Yildizeli Topcu, PhD, Principal Investigator — Trakya University
Locations (1):
- Trakya University Health Science Faculty, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.